CLINICAL TRIAL: NCT02879799
Title: Family Integrated Care (FICare) in Level II NICUs: An Innovative Program for Alberta
Brief Title: Family Integrated Care (FICare) in Level II NICUs
Acronym: FICare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Karen Benzies, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AIHS-PRIHS 201400399
Record Dates: First submitted 2016-05-27; First posted 2016-08-26 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Premature Birth
Keywords: Family-centered care; Family-integrated care; Neonatal intensive care unit; Premature; Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implement Family Integrated Care (Experimental): Dynamic education and support intervention for families of preterm infants.
  Interventions: Other: Implement Family Integrated Care
- Monitor Standard Practices (No Intervention): Standard nursing care of preterm infants and their families.

INTERVENTIONS:
Other: Implement Family Integrated Care — Specially trained FICare nurses will provide education and support for families to provide care for the baby while they are present in the NICU. Study mothers will meet with veteran parents for additional support. Families will keep a log of their activities and costs.
  Arms: Implement Family Integrated Care

SUMMARY:
In Alberta, nearly one in every twelve babies is born too soon (preterm). Preterm babies are at greater risk for breathing and feeding problems, as well as infections, than babies born on their due date (full term). As a result, parents must leave their preterm babies in the hospital to fully develop and become healthy enough to take home. When it is time for discharge, parents are often not ready to look after their baby because they may have limited involvement in the care of their baby in hospital. In addition to the distress and costs to parents of having a baby in hospital, health system costs are also increased the longer a baby is in hospital. The purpose of this project is to test a new way to integrate parents into the care of their baby through a program called Family Integrated Care (FICare). In FICare, parents are educated and supported by nurses to provide care for their baby; nurses and doctors still provide intravenous medications and medical procedures. FICare has been tested in Ontario and shows promise as a better model of care for the small percentage of babies born more than 8 weeks early, who have to spend a long time in hospital.

Now the investigators want to test FICare with the greater percentage of preterm babies who are born 4 to 8 weeks early to see if parents are able to take their baby home sooner, and if their babies are healthier. The investigators also want to know if FICare can reduce distress for parents. The investigators propose to test FICare in Level II Neonatal Intensive Care Units (NICUs) in Alberta by implementing FICare in half the Level II NICUs and comparing the outcomes with the other Level II NICUs who do not use FICare. If FICare improves outcomes for preterm babies and their parents, the investigators will implement it in all Level II NICUs. In Alberta, the investigators want the best quality care for our most vulnerable babies and their parents. This project is aligned with Alberta's Health Research and Innovation Strategy priority of wellness at every age (child and maternal health), and with Alberta Health Services' quality of care goals to increase efficiency, effectiveness, appropriateness, and acceptability of health care services delivery.

DETAILED DESCRIPTION:
Every year, about 15 million of the world's infants are born at <37 weeks gestation (preterm). In Alberta, the preterm birth rate was 8.43% in 2015, representing 4,749 infants. Alberta has the highest rate of preterm birth in Canada, which can be attributed, in part, to delayed child bearing and assisted reproductive technology. Approximately 20% of the earliest (< 32 weeks gestation) and usually the sickest preterm infants require care in a Level III neonatal intensive care unit (NICU). Approximately 80% are moderate to late preterm (32 weeks and zero days [32 0/7] and 36 weeks and six days [36 6/7] gestation; comprising 6.6% of all live births) and require care in a Level II NICU. Compared to their full term counterparts, moderate and late preterm infants are at higher risk for poor health (e.g., increased hospitalizations, respiratory morbidities, and growth and feeding problems) and developmental outcomes, including neurodevelopmental disabilities and cognitive delays, communication and language impairments,] and school-related problems. As gestational age (GA) decreases, the risk of chronic health problems and developmental delays increases. In 2010, care of preterm infants represented the largest category of Alberta's expenditures for pediatric health care at 8.45%, with a total cost of approximately $35 million. The costs associated with preterm infants are greater than for term infants because of increased hospital length of stay (LOS), resource utilization, readmissions, and need for health, education, and social services. Financial consequences for parents of preterm infants are associated with reduced workforce participation and lost earnings, and developmental supports for the infant. Unquantifiable costs are associated with psychological distress, marital distress, and social isolation. Although effective interventions for parents of preterm infants exist, evidence is generally limited to the earliest preterm infants, and cost effectiveness data is lacking. Implementing a new model of care, Family Integrated Care (FICare), in Level II NICUs for moderate to late preterm infants has great potential to improve outcomes of infants and parents, and reduce costs to the health care system and families.

Level II NICUs are a highly technological, critical care environment where healthcare providers (i.e., nurses, physicians, trainees, respiratory therapists, social workers, and others) often unintentionally marginalize parents in the pursuit of optimal care of preterm infants. The unexpected birth of a tiny infant leaves parents in shock, feeling anxious, depressed, isolated, and unprepared to interact with, and care for, their infant. Preterm birth and experiences in the NICU disrupt breastfeeding and the early parent-infant relationship, which is critical for early brain and biological development. The goal of FICare is a change in culture and practice that permits, encourages, and supports parents in their parenting role while their infant is in a Level II NICU. FICare is, in essence, a dynamic educational intervention, with learners (parents), coaches (healthcare providers and veteran NICU parents), curriculum content, and implementation strategies. Veteran parents are those who have had previous experience with their own preterm infant in a Level II NICU. Underpinned by adult learning and change theories, FICare empowers parents to build their knowledge, skill, and confidence so that the family is well-prepared to care for their infant long before discharge. This model is dynamic, whereby parents and healthcare providers openly and mutually negotiate equitable roles during the infant's NICU stay. Thus, roles will change as parents learn to care for their infant.

Philosophically, efforts to keep parents closer to their infant in NICU started in the 1950s with parental presence that permitted visitation in the NICU. Later, family-centred care articulated respect for family in decisions about care. Despite a comprehensive understanding of family-centred care and recognition of its importance, family-centred approaches remain fraught with challenges, including non-facilitative physical space, restrictive access, limited parental involvement in direct infant care, and lack of consistent information. These challenges result in confusion about the parental role in NICU, and leave parents feeling dissatisfied and more like detached visitors than parents. Integrating parents as central to the care of their infant is the next logical step in the evolution of approaches to NICU care.

Existing interventions include skin-to-skin care, psychological support for the parent (primarily mothers), education about the care of a preterm infant, and education of parents as providers of supportive therapy for their infant. A systematic review suggested that psychological support and parenting education showed the greatest effect over the short- (<1 year) and longer- (≥1 year) term. While parenting education can take many forms from simple leaflets with information to self-modeled video interaction guidance, parenting education that actively engages parents with their infant had the greatest impact on parental and infant outcomes. Education that is consistent across care providers is critical to ensure parental belief in the competence of care providers. A positive relationship between parents and providers contributes to increased satisfaction with care, and greater willingness by parents to seek further support for the care of their infant. Further, health care should be individualized to accommodate sequential clinical phases from admission to post-discharge care of the infant.

Adapted from existing family-centred care interventions, the Family Integrated Care (FICare) model was developed and pilot tested with preterm infants ≤ 35 weeks GA in a Level III NICU at Mount Sinai Hospital, Toronto. The pilot study indicates that FICare is feasible and safe in Canada. Compared to 31 matched controls, the 42 infants who received FICare showed increased weight gain and breastfeeding at discharge. FICare reduced LOS by approximately 10% (personal communication, Dr. S. Lee) and mothers reported less stress. Based on these promising results, FICare in Level III NICUs is currently being evaluated in a 19-centre, cRCT; Calgary is a control site. With success in Level III NICUs, Dr. V. Shah (co-investigator) is implementing FICare in four Ontario Level II NICUs. However, the Ontario study is limited by a pre-test/post-test design. Without a randomized controlled train (RCT), evidence of the effectiveness of FICare in Level II NICUs will continue to be plagued by methodological and contextual limitations. The aim of this study is to refine and implement FICare in Level II NICUs across Alberta and evaluate it using a cluster RCT (cRCT).

The investigators hypothesize that compared with standard care, FICare will: (1) decrease LOS (primary outcome); (2) decrease the incidence of nosocomial infections; (3) decrease adverse events (e.g., medication and donor breast milk errors); (4) reduce the number of times infants have feeding suspended (NPO) with concomitant intravenous therapy and/or sepsis workups; (5) reduce readmission and unplanned emergency room and physician visits up to 2 months corrected age (CA); (6) increase parental knowledge, skills, and confidence in caring for their infant at discharge and 2 months CA; (7) increase rates of feeding breast milk and breastfeeding self-efficacy at discharge and 2 months CA; (8) decrease parental psychosocial distress (stress, anxiety, depression) at discharge and 2 months CA, (9) improve healthcare provider satisfaction; and (10) decrease direct and indirect costs because of reduced LOS and readmission.

The FICare Alberta research study was co-developed in collaboration with Alberta Health Services operational leaders and clinicians. Nursing and medical directors at the ten Level II NICUs across Alberta embraced the idea of FICare. Buy-in is particularly notable given that sites were aware that they could be randomized to either FICare or control condition. The investigators addressed the potential for unanticipated compensatory reactions (i.e., demoralization) by offering delayed implementation of FICare at control sites. The investigators discussed development, testing, and execution of the FICare implementation plan, as well as how we can integrate changes for the new model into routine care. The investigators learned that several sites were already using some elements of FICare, albeit in an unstructured and unintegrated way. If results of FICare show improved outcomes and/or reduced costs, we will assist with implementation and provide training to staff at the control sites.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants born between 32 weeks and zero days and 34 weeks and 6 days gestation.
* Mothers of any age who have decision making capacity.
* Mothers who are literate, and speak, read and understand English well enough to provide informed consent, and complete surveys online or via telephone.

Exclusion Criteria:

* Mothers whose infants have serious congenital anomalies that require surgery, or are receiving palliative care.
* Mothers who are not able to communicate in English.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07-26 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Birth admission length of stay | Hospital length of stay in days, expected to range between 14 and 24 days; some infants may require a longer admission
  Time in days from birth (admission) to discharge

SECONDARY OUTCOMES:
Nosocomial infection | From date of birth (admission) to date of discharge from hospital - up to 24 days (may be longer for some infants)
  Number of nosocomial infections from birth (admission) to discharge
Adverse events | From date of birth (admission) to date of discharge from hospital - up to 24 days (may be longer for some infants)
  E.g. medication and breast milk errors
Number of times infant NPO | From date of birth (admission) to date of discharge from hospital - up to 24 days (may be longer for some infants)
  Number of times infant was NPO (nothing by mouth) from birth (admission) to discharge - up to 24 days (may be longer for some infants)
Taking breast milk | On date of admission, date of discharge, and date at 2-months corrected age
  Includes time to full oral feeds from birth
Number of re-admissions to hospital | From date of discharge from hospital to date at 2-months corrected age
Number of emergency room visits | From date of discharge from hospital to date at 2-months corrected age
Number of unplanned visits to physician or other provider | From date of discharge from hospital to date at 2-months corrected age

OTHER OUTCOMES:
Parental confidence in caring for their infant questionnaire | On date of admission, on date of discharge, and at 2-months corrected age
Breastfeeding self-efficacy questionnaire | On date of admission, on date of discharge, and at 2-months corrected age
Parental psychosocial distress (stress, anxiety, depression) questionnaires | On date of admission, date of discharge, and date at 2-months corrected age
Staff satisfaction questionnaire | 12 months post-implementation
Direct industry costs (hospital costs, excluding housekeeping, maintenance, planning and physician times). | From birth admission date to hospital discharge date; from hospital discharge date to 2-months corrected age
Indirect societal costs (out-of-pocket costs to the family including parking, transportation, lodging, food, and time off work) collected in parent journal | From birth admission date to hospital discharge date - up to 24 days (may be longer for some infants)
Demographics (including mother and father age; education; family income; marital status) | Baseline
Maternal health data (including chronic diseases; ART; antenatal steroids; pregnancy complications; mode of delivery; parity/gravida) | Baseline
Infant health data (including DOB; Apgar; multiple birth; admission illness severity; medications; interventions; weight gain) | Date of discharge from hospital - up to 24 days post birth (may be longer for some infants)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Benzies, PhD, Principal Investigator — University of Calgary; Abhay Lodha, MD, Principal Investigator — University of Calgary; Khalid Aziz, MD, Principal Investigator — University of Alberta; Vibhuti Shah, MD, Principal Investigator — University of Toronto
Locations (10):
- Canada (10):
  - Peter Lougheed Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Queen Elizabeth II Hospital, Grande Prairie, Alberta
  - Chinook Regional Hospital, Lethbridge, Alberta
  - Medicine Hat Regional Hospital, Medicine Hat, Alberta
  - Red Deer Regional Hospital, Red Deer, Alberta

IPD SHARING:
Plan to Share IPD: Yes
Negotiations are underway to reposit data with the Alberta Centre for Child, Family and Community Research, Secondary Analyses to Generate Evidence (SAGE)

REFERENCES:
- [Background] March of Dimes, PMNCH, Save the Children, World Health Organization. Born too soon: The global action report on preterm birth. Geneva: World Health Organization; 2012.
- [Background] Alberta Health and Wellness. Interactive Health Data Application, 2015 reproductive health data set. Edmonton, AB: Alberta Health and Wellness, Government of Alberta; 2015. From http://www.ahw.gov.ab.ca/IHDA_Retrieval/selectSubCategory.do
- [Background] Alberta Reproductive Health Report Working Group. Alberta reproductive health: Pregnancies and births table update 2011. Edmonton, AB: Alberta Health and Wellness, Government of Alberta; 2011.
- [Background] Tough SC, Newburn-Cook C, Johnston DW, Svenson LW, Rose S, Belik J. Delayed childbearing and its impact on population rate changes in lower birth weight, multiple birth, and preterm delivery. Pediatrics. 2002 Mar;109(3):399-403. doi: 10.1542/peds.109.3.399. PMID 11875131
- [Background] Tough S, Tofflemire K, Newburn-Cook C, Fraser-Lee N, Benzies K. Increased risks of pregnancy complications and adverse infant outcomes associated with assisted reproduction. International Congress Series; 2004: Elsevier. p. 376-9.
- [Background] Alberta Perinatal Health Program: Provincial Perinatal Report. Alberta Health Services; 2013.
- [Background] Harijan P, Boyle EM. Health outcomes in infancy and childhood of moderate and late preterm infants. Semin Fetal Neonatal Med. 2012 Jun;17(3):159-62. doi: 10.1016/j.siny.2012.02.002. Epub 2012 Mar 13. PMID 22417643
- [Background] Sahni R, Polin RA. Physiologic underpinnings for clinical problems in moderately preterm and late preterm infants. Clin Perinatol. 2013 Dec;40(4):645-63. doi: 10.1016/j.clp.2013.07.012. Epub 2013 Sep 20. PMID 24182953
- [Background] McGowan JE, Alderdice FA, Holmes VA, Johnston L. Early childhood development of late-preterm infants: a systematic review. Pediatrics. 2011 Jun;127(6):1111-24. doi: 10.1542/peds.2010-2257. Epub 2011 May 29. PMID 21624885
- [Background] Johnson S, Evans TA, Draper ES, Field DJ, Manktelow BN, Marlow N, Matthews R, Petrou S, Seaton SE, Smith LK, Boyle EM. Neurodevelopmental outcomes following late and moderate prematurity: a population-based cohort study. Arch Dis Child Fetal Neonatal Ed. 2015 Jul;100(4):F301-8. doi: 10.1136/archdischild-2014-307684. Epub 2015 Apr 1. PMID 25834170
- [Background] Guy A, Seaton SE, Boyle EM, Draper ES, Field DJ, Manktelow BN, Marlow N, Smith LK, Johnson S. Infants born late/moderately preterm are at increased risk for a positive autism screen at 2 years of age. J Pediatr. 2015 Feb;166(2):269-75.e3. doi: 10.1016/j.jpeds.2014.10.053. Epub 2014 Dec 2. PMID 25477165
- [Background] Kerstjens JM, de Winter AF, Bocca-Tjeertes IF, ten Vergert EM, Reijneveld SA, Bos AF. Developmental delay in moderately preterm-born children at school entry. J Pediatr. 2011 Jul;159(1):92-8. doi: 10.1016/j.jpeds.2010.12.041. Epub 2011 Feb 16. PMID 21324481
- [Background] Ballantyne M, Benzies KM, McDonald S, Magill-Evans J, Tough S. Risk of developmental delay: Comparison of late preterm and full term Canadian infants at age 12 months. Early Hum Dev. 2016 Oct;101:27-32. doi: 10.1016/j.earlhumdev.2016.04.004. Epub 2016 Jul 9. PMID 27405053
- [Background] Stene-Larsen K, Brandlistuen RE, Lang AM, Landolt MA, Latal B, Vollrath ME. Communication impairments in early term and late preterm children: a prospective cohort study following children to age 36 months. J Pediatr. 2014 Dec;165(6):1123-8. doi: 10.1016/j.jpeds.2014.08.027. Epub 2014 Sep 23. PMID 25258153
- [Background] Chan E, Quigley MA. School performance at age 7 years in late preterm and early term birth: a cohort study. Arch Dis Child Fetal Neonatal Ed. 2014 Nov;99(6):F451-7. doi: 10.1136/archdischild-2014-306124. Epub 2014 Jun 25. PMID 24966128
- [Background] de Jong M, Verhoeven M, van Baar AL. School outcome, cognitive functioning, and behaviour problems in moderate and late preterm children and adults: a review. Semin Fetal Neonatal Med. 2012 Jun;17(3):163-9. doi: 10.1016/j.siny.2012.02.003. Epub 2012 Feb 23. PMID 22364677
- [Background] van Baar AL, Vermaas J, Knots E, de Kleine MJ, Soons P. Functioning at school age of moderately preterm children born at 32 to 36 weeks' gestational age. Pediatrics. 2009 Jul;124(1):251-7. doi: 10.1542/peds.2008-2315. PMID 19564307
- [Background] Kerstjens JM, de Winter AF, Bocca-Tjeertes IF, Bos AF, Reijneveld SA. Risk of developmental delay increases exponentially as gestational age of preterm infants decreases: a cohort study at age 4 years. Dev Med Child Neurol. 2012 Dec;54(12):1096-101. doi: 10.1111/j.1469-8749.2012.04423.x. Epub 2012 Sep 30. PMID 23020259
- [Background] Schonhaut L, Armijo I, Perez M. Gestational age and developmental risk in moderately and late preterm and early term infants. Pediatrics. 2015 Apr;135(4):e835-41. doi: 10.1542/peds.2014-1957. Epub 2015 Mar 2. PMID 25733752
- [Background] Sun Y, Hsu P, Vestergaard M, Christensen J, Li J, Olsen J. Gestational age, birth weight, and risk for injuries in childhood. Epidemiology. 2010 Sep;21(5):650-7. doi: 10.1097/EDE.0b013e3181e94253. PMID 20585254
- [Background] Dean S. Reporting and analytics. Child Health Strategic Clinical Network meeting. Calgary, AB: Alberta Health Services; 2012, October 12.
- [Background] Petrou S, Khan K. Economic costs associated with moderate and late preterm birth: primary and secondary evidence. Semin Fetal Neonatal Med. 2012 Jun;17(3):170-8. doi: 10.1016/j.siny.2012.02.001. Epub 2012 Feb 23. PMID 22364679
- [Background] Petrou S, Eddama O, Mangham L. A structured review of the recent literature on the economic consequences of preterm birth. Arch Dis Child Fetal Neonatal Ed. 2011 May;96(3):F225-32. doi: 10.1136/adc.2009.161117. Epub 2010 May 20. PMID 20488863
- [Background] Benzies KM, Magill-Evans JE, Hayden KA, Ballantyne M. Key components of early intervention programs for preterm infants and their parents: a systematic review and meta-analysis. BMC Pregnancy Childbirth. 2013;13 Suppl 1(Suppl 1):S10. doi: 10.1186/1471-2393-13-S1-S10. Epub 2013 Jan 31. PMID 23445560
- [Background] Staub K, Baardsnes J, Hebert N, Hebert M, Newell S, Pearce R. Our child is not just a gestational age. A first-hand account of what parents want and need to know before premature birth. Acta Paediatr. 2014 Oct;103(10):1035-8. doi: 10.1111/apa.12716. Epub 2014 Jul 18. No abstract available. PMID 24920539
- [Background] Dayan J, Creveuil C, Marks MN, Conroy S, Herlicoviez M, Dreyfus M, Tordjman S. Prenatal depression, prenatal anxiety, and spontaneous preterm birth: a prospective cohort study among women with early and regular care. Psychosom Med. 2006 Nov-Dec;68(6):938-46. doi: 10.1097/01.psy.0000244025.20549.bd. Epub 2006 Nov 1. PMID 17079701
- [Background] McDonald SW, Benzies KM, Gallant JE, McNeil DA, Dolan SM, Tough SC. A comparison between late preterm and term infants on breastfeeding and maternal mental health. Matern Child Health J. 2013 Oct;17(8):1468-77. doi: 10.1007/s10995-012-1153-1. PMID 23054457
- [Background] Schmucker G, Brisch KH, Kohntop B, Betzler S, Osterle M, Pohlandt F, Pokorny D, Laucht M, Kachele H, Buchheim A. The influence of prematurity, maternal anxiety, and infants' neurobiological risk on mother-infant interactions. Infant Ment Health J. 2005 Sep;26(5):423-441. doi: 10.1002/imhj.20066. PMID 28682494
- [Background] Lasiuk GC, Comeau T, Newburn-Cook C. Unexpected: an interpretive description of parental traumas' associated with preterm birth. BMC Pregnancy Childbirth. 2013;13 Suppl 1(Suppl 1):S13. doi: 10.1186/1471-2393-13-S1-S13. Epub 2013 Jan 31. PMID 23445715
- [Background] Gooding JS, Cooper LG, Blaine AI, Franck LS, Howse JL, Berns SD. Family support and family-centered care in the neonatal intensive care unit: origins, advances, impact. Semin Perinatol. 2011 Feb;35(1):20-8. doi: 10.1053/j.semperi.2010.10.004. PMID 21255703
- [Background] Korja R, Latva R, Lehtonen L. The effects of preterm birth on mother-infant interaction and attachment during the infant's first two years. Acta Obstet Gynecol Scand. 2012 Feb;91(2):164-73. doi: 10.1111/j.1600-0412.2011.01304.x. PMID 22007730
- [Background] Shonkoff JP, Garner AS; Committee on Psychosocial Aspects of Child and Family Health; Committee on Early Childhood, Adoption, and Dependent Care; Section on Developmental and Behavioral Pediatrics. The lifelong effects of early childhood adversity and toxic stress. Pediatrics. 2012 Jan;129(1):e232-46. doi: 10.1542/peds.2011-2663. Epub 2011 Dec 26. PMID 22201156
- [Background] Knowles M. The adult learner: A neglected species. Houston, TX: Gulf Publishing Company; 1973
- [Background] Prochaska JO, DiClemente CC. Transtheoretical therapy: Toward a more integrative model of change. Psychotherapy: Theory, Research & Practice 1982;19:276-88.
- [Background] de Alencar AE, Arraes LC, de Albuquerque EC, Alves JG. Effect of kangaroo mother care on postpartum depression. J Trop Pediatr. 2009 Feb;55(1):36-8. doi: 10.1093/tropej/fmn083. Epub 2008 Dec 9. PMID 19066171
- [Background] Neu M, Robinson J. Maternal holding of preterm infants during the early weeks after birth and dyad interaction at six months. J Obstet Gynecol Neonatal Nurs. 2010 Jul-Aug;39(4):401-14. doi: 10.1111/j.1552-6909.2010.01152.x. PMID 20629927
- [Background] Jefferies AL; Canadian Paediatric Society, Fetus and Newborn Committee. Kangaroo care for the preterm infant and family. Paediatr Child Health. 2012 Mar;17(3):141-6. doi: 10.1093/pch/17.3.141. PMID 23449885
- [Background] Ludington-Hoe SM, Morgan K, Abouelfettoh A. A clinical guideline for implementation of kangaroo care with premature infants of 30 or more weeks' postmenstrual age. Adv. Neonatal Care. 2008;8(3S):S3-S23.
- [Background] Newnham CA, Milgrom J, Skouteris H. Effectiveness of a modified Mother-Infant Transaction Program on outcomes for preterm infants from 3 to 24 months of age. Infant Behav Dev. 2009 Jan;32(1):17-26. doi: 10.1016/j.infbeh.2008.09.004. Epub 2008 Nov 20. PMID 19026450
- [Background] Project AP. Randomised trial of parental support for families with very preterm children. Avon Premature Infant Project. Arch Dis Child Fetal Neonatal Ed. 1998 Jul;79(1):F4-11. doi: 10.1136/fn.79.1.f4. PMID 9797618
- [Background] Ravn IH, Smith L, Lindemann R, Smeby NA, Kyno NM, Bunch EH, Sandvik L. Effect of early intervention on social interaction between mothers and preterm infants at 12 months of age: a randomized controlled trial. Infant Behav Dev. 2011 Apr;34(2):215-25. doi: 10.1016/j.infbeh.2010.11.004. Epub 2011 Mar 2. PMID 21371754
- [Background] Kaaresen PI, Ronning JA, Ulvund SE, Dahl LB. A randomized, controlled trial of the effectiveness of an early-intervention program in reducing parenting stress after preterm birth. Pediatrics. 2006 Jul;118(1):e9-19. doi: 10.1542/peds.2005-1491. PMID 16818541
- [Background] Melnyk BM, Feinstein NF, Alpert-Gillis L, Fairbanks E, Crean HF, Sinkin RA, Stone PW, Small L, Tu X, Gross SJ. Reducing premature infants' length of stay and improving parents' mental health outcomes with the Creating Opportunities for Parent Empowerment (COPE) neonatal intensive care unit program: a randomized, controlled trial. Pediatrics. 2006 Nov;118(5):e1414-27. doi: 10.1542/peds.2005-2580. Epub 2006 Oct 16. PMID 17043133
- [Background] Glazebrook C, Marlow N, Israel C, Croudace T, Johnson S, White IR, Whitelaw A. Randomised trial of a parenting intervention during neonatal intensive care. Arch Dis Child Fetal Neonatal Ed. 2007 Nov;92(6):F438-43. doi: 10.1136/adc.2006.103135. Epub 2007 Feb 14. PMID 17301114
- [Background] Teti DM, Black MM, Viscardi R, et al. Intervention with African American premature infants: Four-month results of an early intervention program. Journal of Early Intervention. 2009;31(2):146-66.
- [Background] Koldewijn K, Wolf MJ, van Wassenaer A, Meijssen D, van Sonderen L, van Baar A, Beelen A, Nollet F, Kok J. The Infant Behavioral Assessment and Intervention Program for very low birth weight infants at 6 months corrected age. J Pediatr. 2009 Jan;154(1):33-38.e2. doi: 10.1016/j.jpeds.2008.07.039. Epub 2008 Sep 10. PMID 18783797
- [Background] Enhancing the outcomes of low-birth-weight, premature infants. A multisite, randomized trial. The Infant Health and Development Program. JAMA. 1990 Jun 13;263(22):3035-42. doi: 10.1001/jama.1990.03440220059030. PMID 2188023
- [Background] Griffin T. Family-centered care in the NICU. J Perinat Neonatal Nurs. 2006 Jan-Mar;20(1):98-102. doi: 10.1097/00005237-200601000-00029. PMID 16508475
- [Background] Van Riper M. Family-provider relationships and well-being in families with preterm infants in the NICU. Heart Lung. 2001 Jan-Feb;30(1):74-84. doi: 10.1067/mhl.2001.110625. PMID 11174370
- [Background] Dunn MS, Reilly MC, Johnston AM, Hoopes RD Jr, Abraham MR. Development and dissemination of potentially better practices for the provision of family-centered care in neonatology: the family-centered care map. Pediatrics. 2006 Nov;118 Suppl 2:S95-107. doi: 10.1542/peds.2006-0913F. PMID 17079629
- [Background] Malusky SK. A concept analysis of family-centered care in the NICU. Neonatal Netw. 2005 Nov-Dec;24(6):25-32. doi: 10.1891/0730-0832.24.6.25. PMID 16383182
- [Background] Dunst CJ, Trivette CM, Hamby DW. Meta-analysis of family-centered helpgiving practices research. Ment Retard Dev Disabil Res Rev. 2007;13(4):370-8. doi: 10.1002/mrdd.20176. PMID 17979208
- [Background] Beck SA, Weis J, Greisen G, Andersen M, Vibeke Z. Room for family-centered care - A qualitative evaluation of a neonatal intensive care unit remodeling project. J. Neonatal Nurs. 2009;15(3):88-99.
- [Background] Cockcroft S. How can family centred care be improved to meet the needs of parents with a premature baby in neonatal intensive care? J. Neonatal Nurs. 2011;18(3):105-10.
- [Background] Newton MS. Family-centered care: current realities in parent participation. Pediatr Nurs. 2000 Mar-Apr;26(2):164-8. PMID 12026270
- [Background] Corlett J, Twycross A. Negotiation of parental roles within family-centred care: a review of the research. J Clin Nurs. 2006 Oct;15(10):1308-16. doi: 10.1111/j.1365-2702.2006.01407.x. PMID 16968435
- [Background] Bracht M, O'Leary L, Lee SK, O'Brien K. Implementing family-integrated care in the NICU: a parent education and support program. Adv Neonatal Care. 2013 Apr;13(2):115-26. doi: 10.1097/ANC.0b013e318285fb5b. PMID 23532031
- [Background] O'Brien K, Bracht M, Macdonell K, McBride T, Robson K, O'Leary L, Christie K, Galarza M, Dicky T, Levin A, Lee SK. A pilot cohort analytic study of Family Integrated Care in a Canadian neonatal intensive care unit. BMC Pregnancy Childbirth. 2013;13 Suppl 1(Suppl 1):S12. doi: 10.1186/1471-2393-13-S1-S12. Epub 2013 Jan 31. PMID 23445639
- [Background] O'Brien K, Bracht M, Robson K, Ye XY, Mirea L, Cruz M, Ng E, Monterrosa L, Soraisham A, Alvaro R, Narvey M, Da Silva O, Lui K, Tarnow-Mordi W, Lee SK. Evaluation of the Family Integrated Care model of neonatal intensive care: a cluster randomized controlled trial in Canada and Australia. BMC Pediatr. 2015 Dec 15;15:210. doi: 10.1186/s12887-015-0527-0. PMID 26671340
- [Derived] Moe AM, Brockway ML, McNeil DA, Afzal AR, Benzies KM. Human milk feeding for moderate and late preterm infants at age 2 months: Insights from a cluster randomized controlled trial 2-month follow-up. PEC Innov. 2024 Sep 19;5:100345. doi: 10.1016/j.pecinn.2024.100345. eCollection 2024 Dec 15. PMID 39391887
- [Derived] Benzies KM, Zanoni P, McNeil DA. Mobilizing strategic inflection points for sustainment of an effective intervention in an integrated learning health system: an interpretive description. Implement Sci Commun. 2024 Sep 30;5(1):106. doi: 10.1186/s43058-024-00644-2. PMID 39350292
- [Derived] Zanoni P, Scime NV, Benzies K, McNeil DA, Mrklas K; Alberta FICare in Level II NICU Study Team; Alberta FICare in Level II NICU Study Team. Facilitators and barriers to implementation of Alberta family integrated care (FICare) in level II neonatal intensive care units: a qualitative process evaluation substudy of a multicentre cluster-randomised controlled trial using the consolidated framework for implementation research. BMJ Open. 2021 Oct 18;11(10):e054938. doi: 10.1136/bmjopen-2021-054938. PMID 34663673
- [Derived] Benzies KM, Aziz K, Shah V, Faris P, Isaranuwatchai W, Scotland J, Larocque J, Mrklas KJ, Naugler C, Stelfox HT, Chari R, Soraisham AS, Akierman AR, Phillipos E, Amin H, Hoch JS, Zanoni P, Kurilova J, Lodha A; Alberta FICare Level II NICU Study Team. Effectiveness of Alberta Family Integrated Care on infant length of stay in level II neonatal intensive care units: a cluster randomized controlled trial. BMC Pediatr. 2020 Nov 28;20(1):535. doi: 10.1186/s12887-020-02438-6. PMID 33246430
- [Derived] Brockway M, Benzies KM, Carr E, Aziz K. Breastfeeding self-efficacy and breastmilk feeding for moderate and late preterm infants in the Family Integrated Care trial: a mixed methods protocol. Int Breastfeed J. 2018 Jul 6;13:29. doi: 10.1186/s13006-018-0168-7. eCollection 2018. PMID 29989087
- [Derived] Benzies KM, Shah V, Aziz K, Isaranuwatchai W, Palacio-Derflingher L, Scotland J, Larocque J, Mrklas K, Suter E, Naugler C, Stelfox HT, Chari R, Lodha A; Alberta FICare Level II NICU Study Team. Family Integrated Care (FICare) in Level II Neonatal Intensive Care Units: study protocol for a cluster randomized controlled trial. Trials. 2017 Oct 10;18(1):467. doi: 10.1186/s13063-017-2181-3. PMID 29017578
- See also: Study Website — http://www.ucalgary.ca/ficare/